CLINICAL TRIAL: NCT07204054
Title: Comparison of Medial Longitudinal Arch Support and Plantar Fascia Stretch Taping Techniques in Plantar Fasciitis
Brief Title: Medial Longitudinal Arch Support and Plantar Fascia Stretch Taping in Plantar Fasciitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/F24C08G30008
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Plantar Fascitis
Keywords: foot function; pain; ankle ROM; arch mobility
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial Longitudinal arch support taping using Low dye Tape (Active Comparator): Medial longitudinal arch support taping is applied using low-dye tape with no tension in the tape; placement of a strip in the area of the metatarsal heads, in the dorsal area placement of a strap on the back, forming a circle with the front strap and in the plantar area; a figure of eight was made, starting from the side of the fifth metatarsal, surrounding the heel and ending at the starting point, the same operation was performed as in point but starting from the hallux. The last part is different, as a strip at the main point of pain, that is, at the insertion towards the medial edge of the foot.
  Ultrasound, stretching and strengthening exercises. Ultrasound will be applied for duration of 7 minutes at the plantar aspect of foot with 1.5 w/cm2 output and continuous mode of frequency of 1MHz. Stretching (5reps with 10 sec hold each stretch) of gastrocnemius and Soleus, toe curl exercise all for a duration of 2 weeks for 2 sessions per week
  Interventions: Other: Medial longitudinal arch support taping using low dye tape
- Fascia Stretch taping using KT tape (Experimental): Fascia Taping which is applied in which In the first step, after the metatarsophalangeal joints were dorsiflexed, the first strap was adhered firmly to the posterior heel at its proximal end. The other end of the strap was cut into four slices of equal width. Each slice was applied with a 50% stretch (50% tensile strain) and attached to the plantar forefoot. In the second step, another strap was applied following the same pattern and overlapped the first strap. In the third step, the last strap was applied with gentle compression across the bases of the four slices beneath the foot and wrapped around the rearfoot.
  Ultrasound, stretching and strengthening exercises. Ultrasound will be applied for duration of 7 minutes at the plantar aspect of foot with 1.5 w/cm2 output and continuous mode of frequency of 1MHz. Stretching (5reps with 10 sec hold each stretch) of gastrocnemius and Soleus and toe curl exercise for a period of twice a week session for 2 weeks
  Interventions: Other: Fascia Stretch taping using KT tape

INTERVENTIONS:
Other: Medial longitudinal arch support taping using low dye tape — Low dye Taping which is applied by patient lying supine on treatment table. No tension is applied due to the characteristics of the tape and it is described in the following steps; placement of a strip in the area of the metatarsal heads, in the dorsal area placement of a strap on the back, forming a circle with the front strap and in the plantar area; a figure of eight was made, starting from the side of the fifth metatarsal, surrounding the heel and ending at the starting point, the same operation was performed as in point but starting from the hallux. The last part is different, as a strip at the main point of pain, that is, at the insertion towards the medial edge of the foot Ultrasound, stretching and strengthening exercises. Ultrasound will be applied for duration of 7 minutes at the plantar aspect of foot with 1.5 w/cm2 output and continuous mode of frequency of 1MHz. Stretching of gastrocnemius and soleus and towel curl exercise.
  Arms: Medial Longitudinal arch support taping using Low dye Tape
Other: Fascia Stretch taping using KT tape — Fascia Taping which is applied in which In the first step, after the metatarsophalangeal joints were dorsiflexed, the first strap was adhered firmly to the posterior heel at its proximal end. The other end of the strap was cut into four slices of equal width. Each slice was applied with a 50% stretch (50% tensile strain) and attached to the plantar forefoot. In the second step, another strap was applied following the same pattern and overlapped the first strap. In the third step, the last strap was applied with gentle compression across the bases of the four slices beneath the foot and wrapped around the rearfoot. Dashed arrows denote the direction of stretch Ultrasound, stretching and strengthening exercises. Ultrasound will be applied for duration of 7 minutes at the plantar aspect of foot with 1.5 w/cm2 output and continuous mode of frequency of 1MHz. Stretching (5reps with 10 sec hold each stretch) of gastrocnemius and Soleus and toe curl exercise
  Arms: Fascia Stretch taping using KT tape

SUMMARY:
Rationale of this research is to evaluate the outcome of two widely used but biomechanically distinct techniques of Taping done for plantar fascia i.e. Fascia taping which supports the fascia, and Low dye taping which realigns with medial longitudinal arch. The significance of this study is to identify which taping technique will improve pain, ankle ROM, foot function and arch flexibility which will help clinicians in identifying the most suitable and effective taping method for the patients

DETAILED DESCRIPTION:
Plantar fasciitis is one of the most common causes of chronic heel pain, leading to reduced mobility, altered gait, and impaired quality of life. Despite its high prevalence, most conventional treatments focus primarily on calf stretching, orthotic devices, or electrotherapy. Taping is a cost effective and powerful treatment technique, this study is being done to identify which taping technique will improve pain, ankle ROM, foot function and arch flexibility in patients with acute and subacute plantar fasciitis. It is a randomized control trial which will be conducted on 36 patient calculated using G* Power software. Participants were randomly assigned to intervention or control group after a baseline assessment using lottery ticket and opaque envelop. All participants in both groups were evaluated on 6 occasions baseline, post-intervention, post every treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants' full filling the criteria given below will be recruited in this study. Diagnosis based on clinical guidelines linked to the International Classiﬁcation of Function, Disability and Health of the Orthopaedic Section of the American Physiotherapy Association.

* Age 25-65 years
* Positive Windlass test
* Tenderness at medial calcaneal tubercle
* Limited ankle dorsiflexion <16
* Acute or subacute stage unilateral plantar fasciitis

Exclusion Criteria:

Individuals with one of the following disorder will be excluded from this study

* Fracture of ankle or foot
* Diabetes
* Neuropathy
* Cognitive impairments/ Psychological disorder
* Rheumatoid Arthritis
* Open wound.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale to assess pain | 2 weeks
  Visual analogue scale to determine the extent of patients pain. The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. VAS has a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best).
Foot Functional index | 2 weeks
  The FFI questionnaire consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week. section (Pain: items 1-9; Disability: 10-18; Activity Limitation: 19-23).
Ankle ROM via Goniometry | 2 weeks
  Using a goniometer to determine the effect on ankle ROM
Arch Height Index and Arch Height flexibility using AHIMS | 2 weeks
  Arch Height Index AHI is the ratio calculated by dividing the height from the floor to the dorsum of the foot by the total foot length. Arch height flexilbility AHF is a change in arch height between sitting and standing positions.
  AHI= Height from floor to dorsum of foot/ Total foot length AHF mm/kN =AH sitting - AH standing/0.4 × body weight

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Bahria Town Stroke and Rehabilitation Centre, Rawalpindi, Punjab Province
  - IIMCT Railway General Hopsital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koh HLA, Lin WH, Kong PW. Comfort and Ground Reaction Forces in Flat-Footed Female Runners: Comparison of Low-Dye Taping versus Sham Taping. J Sports Sci Med. 2020 Aug 13;19(3):620-626. eCollection 2020 Sep. PMID 32874115
- [Background] Garcia-Gomariz C, Hernandez-Guillen D, Nieto-Gil P, Blasco-Garcia C, Alcahuz-Grinan M, Blasco JM. Effects of Kinesiotape versus Low-Dye Tape on Pain and Comfort Measures in Patients with Plantar Fasciitis: A Randomized Clinical Trial. Life (Basel). 2024 Feb 12;14(2):249. doi: 10.3390/life14020249. PMID 38398758
- [Background] Van Tonder T, Allison GT, Hopper D, Grisbrook TL. Multidimensional impact of low-Dye taping on low-load hopping in individuals with and without plantar fasciitis. Phys Ther Sport. 2018 Jan;29:43-49. doi: 10.1016/j.ptsp.2017.11.001. Epub 2017 Nov 8. PMID 29245027
- [Background] Podolsky R, Kalichman L. Taping for plantar fasciitis. J Back Musculoskelet Rehabil. 2015;28(1):1-6. doi: 10.3233/BMR-140485. PMID 24867905